CLINICAL TRIAL: NCT00618930
Title: Moviprep® Versus Fleet Phospho-Soda® (Golden Standard): A Study That Compared Two Laxatives on Patients Undergoing Colo-Rectal Cleansing Prior to an Abdominal Operation.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Piet Pattyn, MD, PhD, University Hospital Ghent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007/320
Record Dates: First submitted 2008-02-06; First posted 2008-02-20 (Estimated); Last update posted 2009-04-15 (Estimated); Status verified 2009-04

CONDITIONS: Colorectal Cleansing Prior Operation
MeSH Terms: interventions — MoviPrep

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Moviprep®
- 2 (Active Comparator): Use of Fleet
  Interventions: Drug: Fleet

INTERVENTIONS:
Drug: Moviprep® — use of Moviprep®
  Arms: 1
Drug: Fleet — Use of Fleet
  Arms: 2

SUMMARY:
The patients are assigned by randomisation on one of the two laxatives. After cleansing they have to fill in an evaluation form to report their findings and difficulties. Also the surgeon will be asked to fill in a score-form to report all details concerning the bowel preparation.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Older than 18
* Informed consent signed
* Mode of surgery

Exclusion Criteria:

* Renal disease
* Heart failure
* Dehydration
* Abdominal obstruction
* Abdominal perforation
* Abdominal paralysis
* Toxic megacolon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-02; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
colorectal cleansing | prior operation

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be